CLINICAL TRIAL: NCT02741284
Title: Oxygen for Category II Intrauterine Fetal Resuscitation: A Randomized, Noninferiority Trial
Brief Title: Oxygen for Intrauterine Resuscitation of Category II Fetal Heart Tracings
Acronym: O2C2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201602164
Record Dates: First submitted 2016-04-10; First posted 2016-04-18 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Electronic Fetal Monitoring; Fetal Hypoxia; Fetal-Placental Circulation
MeSH Terms: conditions — Fetal Hypoxia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Oxygen (Experimental): Room air
  Interventions: Drug: Room air
- Oxygen (Active Comparator): 10L oxygen by nonrebreather mask
  Interventions: Drug: 10L Oxygen by nonrebreather mask

INTERVENTIONS:
Drug: Room air
  Arms: No Oxygen
Drug: 10L Oxygen by nonrebreather mask
  Arms: Oxygen

SUMMARY:
Maternal oxygen administration for concerning fetal heart rate tracing (FHT) patterns is common practice on Labor and Delivery units in the United States. Despite the broad use of oxygen, it is unclear if this practice is beneficial for the fetus. The purpose of this study is to compare oxygen to room air in patients with Category II fetal heart tracings with regard to neonatal acid-base status, subsequent tracings, and production of reactive oxygen species

DETAILED DESCRIPTION:
Maternal oxygen administration for concerning fetal heart rate tracing (FHT) patterns is common practice on Labor and Delivery units in the United States. Despite the broad use of oxygen, it is unclear if this practice is beneficial for the fetus. Category II FHT, as defined by the National Institute of Child Health and Human Development (NICHD) (Robinson), is a broad class of FHT patterns that may suggest cord compression and/or placental insufficiency for which oxygen is most commonly administered. Although some animal and human studies (Khazin, Althabe) have demonstrated that maternal hyperoxygenation can alleviate such fetal heart rate decelerations, this purported benefit has not been shown to translate into improved fetal outcomes, particularly in relation to acid-base status. In fact, some studies suggest harm with oxygen use due to lower umbilical artery pH and increased delivery room resuscitation (Nesterenko, Thorp) or increased free radical activity (Khaw). Given the indeterminate evidence for this ubiquitously employed resuscitation technique, there is an urgent need to further study the utility of maternal oxygen administration in labor for fetal benefit.

We propose a randomized controlled non-inferiority trial comparing oxygen to room air in patients with Category II FHT. Our central hypothesis is that room air alone is not inferior to oxygen administration with regard to neonatal acid-base status and FHT and may in fact, be a safer option for resuscitation due to less production of reactive oxygen species.

Primary Aim: Determine the effect of maternal oxygen administration for Category II FHT on arterial umbilical cord lactate.

Hypothesis: Room air, as a substitute for oxygen supplementation, is no different than oxygen in altering the acid-base status of the neonate as reflected in umbilical arterial (UA) lactate.

Fetal hypo-oxygenation, as reflected by decelerations in the FHT, results in metabolic acidosis due to a shift from aerobic to anaerobic metabolism in which lactate and hydrogen ion production significantly increase causing a decrease in pH (Tuuli). Elevated umbilical cord lactate has been shown to be a surrogate for fetal metabolic acidosis and resultant neonatal morbidity (Tuuli, Westgren). The theorized benefit of maternal oxygen administration is increased oxygen delivery to the fetus resulting in reversal of anaerobic metabolism/ metabolic acidosis. This, however, has not been substantiated by evidence thus far. Women with persistent Category II FHT tracing will be randomly assigned to supplemental oxygen or room air. The primary outcome will be umbilical arterial lactate level, and secondary outcomes will be other umbilical cord gas parameters including UA pH, UV oxygen saturation, and UA base deficit.

Secondary Aim #1: Characterize the effect of oxygen administration on fetal heart tracing patterns Hypothesis: Oxygen administration will be associated with a rate of persistent Category II FHT that is not different from those exposed to room air.

Oxygen is typically administered as a response to FHT interpretation. Evidence thus far shows that Category II FHT are associated with a wide spectrum of neonatal outcomes and therefore do not uniformly reflect fetal acid-base status (Cahill, Frey). Hence, evaluating the effect of oxygen on subsequent FHT categorization is pivotal to labor management. The outcome that will be investigated is rate of persistent Category II FHT after intervention.

Secondary Aim #2: Evaluate the safety of oxygen administration by measuring reactive oxygen species (ROS) in maternal and neonatal blood.

Hypothesis: Oxygen administration will be associated with increased oxidative stress in maternal and neonatal cord blood as represented by malondialdehyde (MDA).

Over-oxygenation can result in free radical or ROS formation that have detrimental downstream effects. The presence of reactive oxygen species results in degradation of lipids in the cell membrane and resultant formation of malondialdehyde (MDA) (Dalle-Donne), which has been studied as a surrogate for oxidative stress (Ilhan, Pryor, Suhail, Lorente).

This study will be a prospective, randomized non inferiority trial to be conducted a single center. This study will include term, singleton patients admitted to Labor& Delivery for spontaneous labor or labor induction. Multiples, significant fetal anomalies, Category III FHT, umbilical artery doppler abnormalities and preterm pregnancies will be excluded. Additionally, women will be excluded if oxygen is required for maternal indications such as hypooxygenation or cardiopulmonary disease. Our primary objective will be umbilical cord lactate. Secondary objectives include additional cord gas parameters including umbilical artery pH, umbilical artery base deficit, and umbilical vein oxygen saturation; FHT categorization and deceleration patterns; maternal and umbilical cord blood measurement of malondialdehyde. Women will be consented at time of admission for labor and randomized when at least 6cm dilated with Category II FHT necessitating provider intervention.

ELIGIBILITY:
Inclusion Criteria:

* Term, singleton patients admitted to Labor& Delivery for spontaneous labor or labor induction

Exclusion Criteria:

* Multiple pregnancy
* Significant fetal anomalies
* Category III FHT
* Umbilical artery doppler abnormalities
* Maternal hypooxygenation or need for oxygen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Robinson B, Nelson L. A Review of the Proceedings from the 2008 NICHD Workshop on Standardized Nomenclature for Cardiotocography: Update on Definitions, Interpretative Systems With Management Strategies, and Research Priorities in Relation to Intrapartum Electronic Fetal Monitoring. Rev Obstet Gynecol. 2008 Fall;1(4):186-92. PMID 19173023
- [Background] Khazin AF, Hon EH, Hehre FW. Effects of maternal hyperoxia on the fetus. I. Oxygen tension. Am J Obstet Gynecol. 1971 Feb 15;109(4):628-37. doi: 10.1016/0002-9378(71)90639-9. No abstract available. PMID 5100084
- [Background] Althabe O Jr, Schwarcz RL, Pose SV, Escarcena L, Caldeyro-Barcia R. Effects on fetal heart rate and fetal pO2 of oxygen administration to the mother. Am J Obstet Gynecol. 1967 Jul 15;98(6):858-70. doi: 10.1016/0002-9378(67)90205-0. No abstract available. PMID 6027716
- [Background] Thorp JA, Trobough T, Evans R, Hedrick J, Yeast JD. The effect of maternal oxygen administration during the second stage of labor on umbilical cord blood gas values: a randomized controlled prospective trial. Am J Obstet Gynecol. 1995 Feb;172(2 Pt 1):465-74. doi: 10.1016/0002-9378(95)90558-8. PMID 7856671
- [Background] Nesterenko TH, Acun C, Mohamed MA, Mohamed AN, Karcher D, Larsen J Jr, Aly H. Is it a safe practice to administer oxygen during uncomplicated delivery: a randomized controlled trial? Early Hum Dev. 2012 Aug;88(8):677-81. doi: 10.1016/j.earlhumdev.2012.02.007. Epub 2012 Mar 23. PMID 22445187
- [Background] Khaw KS, Wang CC, Ngan Kee WD, Pang CP, Rogers MS. Effects of high inspired oxygen fraction during elective caesarean section under spinal anaesthesia on maternal and fetal oxygenation and lipid peroxidation. Br J Anaesth. 2002 Jan;88(1):18-23. doi: 10.1093/bja/88.1.18. PMID 11883375
- [Background] Tuuli MG, Stout MJ, Shanks A, Odibo AO, Macones GA, Cahill AG. Umbilical cord arterial lactate compared with pH for predicting neonatal morbidity at term. Obstet Gynecol. 2014 Oct;124(4):756-761. doi: 10.1097/AOG.0000000000000466. PMID 25198278
- [Background] Westgren M, Divon M, Horal M, Ingemarsson I, Kublickas M, Shimojo N, Nordstrom L. Routine measurements of umbilical artery lactate levels in the prediction of perinatal outcome. Am J Obstet Gynecol. 1995 Nov;173(5):1416-22. doi: 10.1016/0002-9378(95)90627-4. PMID 7503179
- [Background] Cahill AG, Roehl KA, Odibo AO, Macones GA. Association and prediction of neonatal acidemia. Am J Obstet Gynecol. 2012 Sep;207(3):206.e1-8. doi: 10.1016/j.ajog.2012.06.046. PMID 22939728
- [Background] Frey HA, Tuuli MG, Shanks AL, Macones GA, Cahill AG. Interpreting category II fetal heart rate tracings: does meconium matter? Am J Obstet Gynecol. 2014 Dec;211(6):644.e1-8. doi: 10.1016/j.ajog.2014.06.033. Epub 2014 Jun 17. PMID 24949543
- [Background] Dalle-Donne I, Rossi R, Colombo R, Giustarini D, Milzani A. Biomarkers of oxidative damage in human disease. Clin Chem. 2006 Apr;52(4):601-23. doi: 10.1373/clinchem.2005.061408. Epub 2006 Feb 16. PMID 16484333
- [Background] Ilhan N, Ilhan N, Simsek M. The changes of trace elements, malondialdehyde levels and superoxide dismutase activities in pregnancy with or without preeclampsia. Clin Biochem. 2002 Jul;35(5):393-7. doi: 10.1016/s0009-9120(02)00336-3. PMID 12270770
- [Background] Pryor WA, Stanley JP. Letter: A suggested mechanism for the production of malonaldehyde during the autoxidation of polyunsaturated fatty acids. Nonenzymatic production of prostaglandin endoperoxides during autoxidation. J Org Chem. 1975 Nov 28;40(24):3615-7. doi: 10.1021/jo00912a038. No abstract available. PMID 1185332
- [Background] Suhail M, Suhail S, Gupta BK, Bharat V. Malondialdehyde and Antioxidant Enzymes in Maternal and Cord Blood, and their Correlation in Normotensive and Preeclamptic Women. J Clin Med Res. 2009 Aug;1(3):150-7. doi: 10.4021/jocmr2009.07.1252. Epub 2009 Aug 12. PMID 22493649
- [Background] Lorente L, Martin MM, Abreu-Gonzalez P, Dominguez-Rodriguez A, Labarta L, Diaz C, Sole-Violan J, Ferreres J, Cabrera J, Igeno JC, Jimenez A. Sustained high serum malondialdehyde levels are associated with severity and mortality in septic patients. Crit Care. 2013 Dec 11;17(6):R290. doi: 10.1186/cc13155. PMID 24326199
- [Background] Lorente L, Martin MM, Abreu-Gonzalez P, Ramos L, Argueso M, Caceres JJ, Sole-Violan J, Lorenzo JM, Molina I, Jimenez A. Association between serum malondialdehyde levels and mortality in patients with severe brain trauma injury. J Neurotrauma. 2015 Jan 1;32(1):1-6. doi: 10.1089/neu.2014.3456. PMID 25054973
- [Derived] Raghuraman N, Wan L, Temming LA, Woolfolk C, Macones GA, Tuuli MG, Cahill AG. Effect of Oxygen vs Room Air on Intrauterine Fetal Resuscitation: A Randomized Noninferiority Clinical Trial. JAMA Pediatr. 2018 Sep 1;172(9):818-823. doi: 10.1001/jamapediatrics.2018.1208. PMID 30039159

RESULTS

PARTICIPANT FLOW:
Groups:
- Room Air: Room air, no mask
Period: Overall Study
Arm/Group | Room Air | Oxygen
Started | 57 | 57
Completed | 51 | 48
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only compared in all patients included in the final analysis. (Randomized patients without paired umbilical cord gases were excluded from this analysis, as the primary outcome required paired cord gases). 48 out of 57 in oxygne and 51 out of 57 in room air had paired gases.
Groups:
- Total: Total of all reporting groups
Arm/Group | Room Air | Oxygen | Total
Number analyzed (Participants) | 51 | 48 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (5.3) | 27.3 (6.3) | 27.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 99
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Baseline characteristics were only compared in patients with paired umbilical cord gases (51 in room air group, and 48 in oxygen group)
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 3 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 40 | 36 | 76
    White | 10 | 8 | 18
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.7 (7.3) | 26.9 (6.5) | 27.3 (6.9)
Gestational age at delivery [Mean (Standard Deviation); unit: weeks] | 39.1 (1.1) | 39.2 (1.1) | 39.1 (1.1)
Nulliparity [Count of Participants; unit: Participants] | 6 | 5 | 11
Chronic hypertension [Count of Participants; unit: Participants] | 6 | 3 | 9
Preeclampsia [Count of Participants; unit: Participants] | 3 | 0 | 3
Pregestational diabetes [Count of Participants; unit: Participants] | 0 | 0 | 0
Tobacco use [Count of Participants; unit: Participants] | 8 | 6 | 14
Illicit drug use [Count of Participants; unit: Participants] | 8 | 12 | 20
Alcohol [Count of Participants; unit: Participants] | 2 | 0 | 2
Induction of labor [Count of Participants; unit: Participants] | 36 | 34 | 70
Oxytocin [Count of Participants; unit: Participants] | 45 | 43 | 88
Chorioamnionitis [Count of Participants; unit: Participants] | 0 | 0 | 0
Epidural [Count of Participants; unit: Participants] | 50 | 44 | 94
Hematocrit on admission [Mean (Standard Deviation); unit: Percentage of red blood cells] | 32.5 (3.2) | 32.8 (3.5) | 32.6 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Umbilical Artery Lactate at Delivery
Description: Determined by umbilical artery cord gas collected at time of delivery and only in patients with paired (umbilical artery and umbilical vein) cord gases.
Time Frame: At delivery
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 51 | 48
mmol/L | 3.5 [3.1 to 4.0] | 3.4 [3.0 to 3.8]
Statistical Analysis 1: Comparison: Room Air vs Oxygen; Test type: Non-Inferiority — A noninferiority margin of 30% (mean difference <1.0 mmol/l) was pre-specified as it corresponds to an upper umbilical artery lactate cut-off value of 4.5 mmol/L, above which there is an increased risk of neonatal morbidity; p = 0.69, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.5 to 0.7]

2. Secondary Outcome: Umbilical Artery pH
Description: as for outcome 1
Time Frame: At time of delivery
Measure: Mean (95% Confidence Interval); unit: pH units
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 51 | 48
pH units | 7.26 [7.24 to 7.28] | 7.25 [7.23 to 7.27]
Statistical Analysis 1: Comparison: Room Air vs Oxygen; pH; Test type: Non-Inferiority — Noninferiority margin 30%; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.01 to 0.03]

3. Secondary Outcome: Mode of Delivery
Description: Delivery via Cesarean section, operative vaginal delivery (forceps or vacuum), or spontaneous vaginal delivery
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 51 | 48
Participants
  Cesarean delivery | 2 | 6
  Cesarean delivery for non reassuring fetal status | 0 | 2
  Operative vaginal delivery | 6 | 1
  Spontaenous vaginal delivery | 43 | 41
Statistical Analysis 1: Comparison: Room Air vs Oxygen; Cesarean delivery; Test type: Superiority; p < 0.05, Chi-squared; Risk Ratio (RR) = 0.32, 95% CI 2-sided [0.07 to 1.48]
Statistical Analysis 2: Comparison: Room Air vs Oxygen; Cesarean delivery for non reassuring fetal status; Test type: Superiority; p < 0.05, Chi-squared; Risk Ratio (RR) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 3: Comparison: Room Air vs Oxygen; Operative vaginal delivery; Test type: Superiority; p < 0.05, Chi-squared; Risk Ratio (RR) = 5.65, 95% CI 2-sided [0.71 to 45.20]

4. Secondary Outcome: Umbilical Artery pCO2
Description: Partial pressure of carbon dioxide as collected on cord gases at time of delivery
Time Frame: At time of delivery
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 51 | 48
mmHg | 55.9 [53.5 to 58.2] | 57.4 [54.2 to 60.6]
Statistical Analysis 1: Comparison: Room Air vs Oxygen; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Net) = -1.5, 95% CI 2-sided [-5.4 to 2.4]

5. Secondary Outcome: Umbilical Artery pO2
Description: Partial pressure of oxygen as collected on cord gases at time of delivery
Time Frame: Time of delivery
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 51 | 48
mm Hg | 19.7 [17.5 to 22.0] | 24.4 [20.0 to 28.8]
Statistical Analysis 1: Comparison: Room Air vs Oxygen; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Net) = -4.7, 95% CI 2-sided [-9.6 to 0.1]

6. Secondary Outcome: Umbilical Artery Base Deficit
Description: As determined by cord gas collection at time of delivery
Time Frame: At time of delivery
Measure: Mean (95% Confidence Interval); unit: meq/L
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 51 | 48
meq/L | -3.6 [-4.3 to -2.9] | -3.6 [-4.3 to -2.9]
Statistical Analysis 1: Comparison: Room Air vs Oxygen; Test type: Superiority; p = 0.99, t-test, 2 sided; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.0 to 1.0]

7. Other Pre Specified Outcome: Number of Patients With Resolved Recurrent Decelerations
Description: Number of patients with resolution of recurrent variable or recurrent late decelerations within 60 minutes of randomization
Time Frame: 60 minutes after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | No Oxygen | Oxygen
Number analyzed (Participants) | 57 | 57
Participants | 49 | 43

ADVERSE EVENTS:
Time Frame: Until neonate was discharged from hospital. (Up to 1 month after delivery)
Description: Does not differ from clinicaltrials.gov definitions
Arm/Group | Room Air | Oxygen
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT02741284/Prot_SAP_000.pdf